CLINICAL TRIAL: NCT02276131
Title: Human Factors and Home Use Study of the Vigilant Diabetes Management Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSpark Technologies, Inc. (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: VG1HFHUS1
Record Dates: First submitted 2014-10-20; First posted 2014-10-28 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usability testing (Experimental): Patients will participate in summative human factors testing of the Vigilant Diabetes Management Application in a controlled environment and during home use testing. Clinicians will participate in summative human factors testing in a controlled environment.
  Interventions: Device: Vigilant Diabetes Management Application

INTERVENTIONS:
Device: Vigilant Diabetes Management Application — Human factors and usability assessment of the device in the hands of diabetes subjects and caregivers

SUMMARY:
A human factors and home use study to assess whether subjects with diabetes and their caregivers can understand feedback received from the Vigilant Diabetes Management Application about their blood glucose patterns and whether the decisions made in response to device feedback are made in accordance with the intended use.

ELIGIBILITY:
Inclusion Criteria:

* Persons with diabetes mellitus testing blood glucose 3 or more times per day
* Clinicians who see diabetes patients

Exclusion Criteria:

* Admission for diabetic ketoacidosis in the 6 months prior to enrollment
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
* Patients who are not willing to share their glucose meter data, or do not perform the tasks asked of them and follow instructions for the study will be excluded
* Pregnancy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adequate understanding of algorithmic feedback based on surveyed responses (Measure: units on a scale) | 1 month home use
  An exit questionnaire will survey participants about comprehension of algorithmic feedback. Across all 5-point rating scales, the average rating will be determined.
Successful completion of frequent and risk-related tasks (Measure: Percent of tasks successfully completed) | Controlled in-office testing for up to 2 hours
  Percent successful initial or reattempt task completion across the range of usability tasks. Example: One task is to access the "Trends" screen to review and interpret weekly and monthly trend data for blood glucose variability and average glucose values.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Anderson, MD, Principal Investigator — University of Virginia